CLINICAL TRIAL: NCT06048458
Title: Cancer Treatment Related Cardiovascular Toxicity: Comprehensive Myocardial and Vascular Phenotyping
Acronym: PC-TOX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 142669
Record Dates: First submitted 2022-04-27; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-12

CONDITIONS: Cardiovascular Diseases; Cardiotoxicity; Fluorouracil Adverse Reaction; Malignancy; Colorectal Cancer; Oesophagus Cancer; Gastric Cancer; Pancreatic Cancer
Keywords: Cardio-oncology; Cardiotoxicity; Fluoropyrimidine cardiotoxicity
MeSH Terms: conditions — Cardiovascular Diseases; Cardiotoxicity; Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Stable patients with gastrointestinal malignancies will be recruited to this 3 timepoint study prior to initiation of fluoropyrimidine chemotherapy. All investigations will be performed at baseline, at the end of cycle 1 and 4-6 weeks post completion of treatment.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance with stress perfusion; Diagnostic Test: CT coronary angiography; Diagnostic Test: Retinal OCT angiography; Diagnostic Test: Sublingual microscopy (GlycoCheck); Diagnostic Test: Serum cardiac biomarkers (High sensitivity troponin, NT pro BNP)
- Cohort 2: Patients with gastrointestinal malignancies presenting to hospital with acute symptoms of fluoropyrimidine cardiotoxicity. All investigations will be performed during the acute presentation and the second visit will be performed 4-6 weeks post completion of treatment.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance with stress perfusion; Diagnostic Test: CT coronary angiography; Diagnostic Test: Retinal OCT angiography; Diagnostic Test: Sublingual microscopy (GlycoCheck); Diagnostic Test: Serum cardiac biomarkers (High sensitivity troponin, NT pro BNP)

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance with stress perfusion — Cardiac MRI scan to assess changes in left ventricular function, parametric mapping, strain and myocardial blood flow. In cohort 1 this will be performed pre, during and on completion of treatment. In cohort 2 this will be performed during the acute presentation and on completion of treatment.
Diagnostic Test: CT coronary angiography — CT coronary angiogram at baseline only in both cohorts to assess for coronary artery disease
Diagnostic Test: Retinal OCT angiography — Retinal OCTa to assess changes in retinal vasculature. In cohort 1 this will be performed pre, during and on completion of treatment. In cohort 2 this will be performed during the acute presentation and on completion of treatment.
Diagnostic Test: Sublingual microscopy (GlycoCheck) — To determine changes in sublingual microvascular health. In cohort 1 this will be performed pre, during and on completion of treatment. In cohort 2 this will be performed during the acute presentation and on completion of treatment.
Diagnostic Test: Serum cardiac biomarkers (High sensitivity troponin, NT pro BNP) — Performed to assess for myocardial injury. In cohort 1 this will be performed pre, during and on completion of treatment. In cohort 2 this will be performed during the acute presentation and on completion of treatment.

SUMMARY:
Observational prospective cohort study designed to assess the mechanisms of fluoropyrimidine induced cardiovascular toxicity.

DETAILED DESCRIPTION:
Fluoropyrimidine (5-FU and Capecitabine) based chemotherapy regimens form the cornerstone of treatments for gastrointestinal (GI) cancers. Fluoropyrimidines however, are associated with the development of cardiovascular toxicity which can take on different forms including chest pain, myocardial infarction, arrhythmias, heart failure and sudden death. The underlying mechanisms of cardiovascular toxicity are not fully understood.

The investigators will use quantitative cardiovascular magnetic resonance perfusion imaging, CT coronary angiography, extra-cardiac vascular assessments and serum cardiac biomarkers to improve insights into the pathophysiology of fluoropyrimidine cardiotoxicity. All enrolled participants in this two centre study will have GI cancers requiring treatment with fluoropyrimidine chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Gastrointestinal malignancy
* Receiving fluoropyrimidine chemotherapy

Exclusion Criteria:

* Participants unable or unwilling to provide consent
* Participants that have a conventional contraindication for magnetic resonance imaging (MRI) including permanent implantable cardiac devices, ferromagnetic implants, pregnancy, large body size not fitting into the scanner bore and severe claustrophobia will be excluded
* Participants that have a conventional contraindication for adenosine stress perfusion including a history of trifascicular block or of second-degree heart block or higher on ECG, or uncontrolled asthma.
* Participants with significant renal impairment (eGFR<30ml/min)
* History of allergy to adenosine, gadolinium or iodinated contrast
* Patients with terminal illness (life expectancy <6 months) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with gastrointestinal malignancies being treated with a fluoropyrimidine based chemotherapy regimen.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial blood flow from baseline with adenosine stress assessed by quantitative perfusion cardiac MRI | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction from baseline | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in left ventricular extracellular volume from baseline | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in left ventricular global longitudinal strain from baseline | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in N-terminal pro B-type natriuretic peptide (NT-pro BNP) | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in high sensitivity troponin T | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in sublingual perfused boundary region | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in sublingual capillary density | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment
Change in retinal vessel density | 6 months
  Assessed at baseline, following cycle 1 and 4-6 weeks post completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Manisty, PhD, Principal Investigator — UCL
Locations (1):
- St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No